CLINICAL TRIAL: NCT02189005
Title: A Prospective, Double Blind, Placebo-Controlled, Randomized, Multicentric, Study to Evaluate the Efficacy and Safety of PreCrea®, a Twice-daily Dietary Supplement in People With Higher Than Normal Blood Sugar Levels.
Brief Title: Study to Evaluate Safety and Efficacy of PreCrea® on Subjects With Higher Than Normal Blood Sugar Levels
Acronym: Precrea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Joe Fenn (Industry)
Responsible Party: Sponsor-Investigator, Joe Fenn, Sponsor-Medical Director, PreEmptive Meds, Pvt. Ltd
Organization: PreEmptive Meds, Pvt. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Precre/Nutra001/PMI13
Record Dates: First submitted 2014-07-11; First posted 2014-07-14 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus; Pre-Diabetes; Hyperglycemia; Metabolic Syndrome
Keywords: High blood sugar; High HbA1C; hyperglycemia; Pre-Diabetes; Natural Supplement for Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Hyperglycemia; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PreCrea (Experimental): Study dietary supplement (Precrea 600 mg capsules) will be given to subjects twice daily 30 mins before food for 90 days along with life style modification program.
  Interventions: Dietary Supplement: Study dietary supplement (PreCrea 600 mg capsules)
- Placebo 600 mg capsules (Placebo Comparator): Placebo was given to patients twice daily 30 mins before food for 90 days along with lifestyle modification program.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Study dietary supplement (PreCrea 600 mg capsules) — Study dietary supplement (PreCrea 600 mg capsules) will be given to subjects twice daily 30 mins before food for 90 days along with life style modification.
  Other Names: PreCrea, Natural Sugar Lowerig Supplement, Predisease
  Arms: PreCrea
Dietary Supplement: Placebo
  Other Names: Placebo 600mg capsules
  Arms: Placebo 600 mg capsules

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of PreCrea® on subjects with higher than normal blood sugar levels.

DETAILED DESCRIPTION:
A Prospective, Double Blind, Placebo-Controlled, Randomized, Multicentric, study to evaluate the efficacy and safety of PreCrea®, a twice-daily dietary supplement in people with higher than normal blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years to ≤ 65 years
2. Newly diagnosed Male or Female participants with higher than normal blood sugar levels (FPG >100 mg/dL) on of Pre-Diabetes and Diabetes Mellitus during screening and not on any treatment
3. Ability to understand and willingness to sign and date a written Informed Consent Document at the screening visit before any protocol- specific procedures are performed and willing to adhere to the protocol and entire trial procedures

Exclusion Criteria:

1. Subjects with Type 1 Diabetes Mellitus
2. Participants on insulin therapy and other oral anti-diabetic agents or having uncontrolled diabetes.
3. Stroke, myocardial infarction, coronary artery bypass graft (CABG) percutaneous transluminal coronary angioplasty (PTCA) or angina pectoris within the last 12 months.
4. Cardiac status New York Heart Association class III-IV
5. Uncontrolled blood pressure > 150 mmhg systolic and > 100 mmhg diastolic
6. Impaired renal function as shown by but not limited to serum creatinine ≥ 1.5 mg/dl for males and ≥ 1.4 mg/dl for female
7. Clinically significant peripheral edema
8. Clinical evidence of active liver disease or serum alenine aminotransferase (ALT) or aspartate amino transferase (AST) 2.5 times the upper limit of the normal range (2.5 X ULN)
9. Participants on steroid
10. Pregnancy or lactating women
11. Known hypersensitivity to any of the study drugs
12. Any malignancy within the last 5 years, with exception of adequately treated basal or squamous cell carcinoma of the skin or adequately treated carcinoma insitu.
13. Current addiction or current alcohol abuse or history of substance or alcohol abuse within the last 2 years
14. Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
15. Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study. Subject unlikely to comply with protocol e.g. uncooperative attitude, inability to return for follow up visits and unlikelihood completing of the study.
16. Any disease or condition that in the opinion of the investigator and/or sponsor may interfere with the completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of Dietary Supplement PreCrea 600 mg twice-daily in lowering Hemoglobin A1c (Hb A1c) levels | Day 1(Baseline) to Day 90 (End of Study)
  Change in HbA1c % from baseline (Day 1) to end of supplementation/treatment after 90 days
Safety of Dietary Supplement PreCrea 600 mg twice-daily | Day 1 (Baseline) to Day 90 (End of Study)
  Measure changes in Renal Function Tests: Blood Urea Nitrogen (BUN) from baseline (Day 1) to end of study (Day 90); Serum Creatinine from baseline (Day 1) to end of study (Day 90)

SECONDARY OUTCOMES:
Efficacy of Dietary Supplement PreCrea 600 mg twice-daily in lowering Fasting Plasma Glucose (FPG) | Day 1 (Baseline) to Day 90 (End of Study)
  Change in FPG % from baseline (Day1) to end of supplementation/treatment after 90 days

OTHER OUTCOMES:
Safety of Dietary Supplement PreCrea 600 mg twice-daily with Liver Function | Baseline (Day 1) to End of Study (Day 90)
  Measure changes in Liver Function Tests: Aspartate Aminotransferase (AST) from baseline (Day 1) to End of Study (Day 90); Alanine Aminotransferase (ALT) from baseline (Day1) to End of Study (Day 90); Alkanine Phosphatase (ALP) from baseline (Day1) to End of Study (Day 90

CONTACTS AND LOCATIONS:
Locations (6):
- India (6):
  - Dia Care- Diabetes Care and Hormone Clinic, Ahmedabad, Gujarat
  - St. Johns College and Hospital, Bangalore, Karnataka
  - Totall Diabetes and Hormone Institution, Indore, Madhya Pradesh
  - Bhatia Hospital, Mumbai, Maharashtra
  - Inamdar Multispeciality Hospital, Pune, Maharashtra
  - Diabetes Care Centre, Jaipur, Rajasthan